CLINICAL TRIAL: NCT03910946
Title: Prevalence of Latent Tuberculosis in High Risk Children Attending Pediatric Hospital of Assiut University
Brief Title: Prevalence of Latent Tuberculosis in High Risk Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, nasef safwat lemby, doctor, Assiut University
Other Study IDs: latent tuberculosis
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis | interventions — Tuberculin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetic and renal: all cases included in the study will be subjected to : Full clinical history to rule out active TB ( history of current prolonged cough, haemoptysis, fever, night sweats, weight loss, chest pain, shortness of breath, fatigue.) Chest x ray TST (tuberculin sensitivity test) : injecting a 0.1 mL of liquid containing 5 TU (tuberculin units) PPD (purified protein derivative) into the top layers of skin of the forearm and read skin tests 48-72 hours after the injection
  Interventions: Drug: Tuberculin, Purified Protein 5Unt/0.1 mL Solution

INTERVENTIONS:
Drug: Tuberculin, Purified Protein 5Unt/0.1 mL Solution — Tuberculosis (diagnosis)-Tuberculin, purified protein derivative (PPD) is indicated as a diagnostic aid in the detection of Mycobacterium tuberculosis infection. It is also indicated when BCG vaccination or isoniazid prophylaxis is being considered
  Other Names: mantoux test

SUMMARY:
identify the prevalence of latent tuberculosis (according to new guideline ;NICE tuberculosis) among these high risk groups of children and notify ministry of health

DETAILED DESCRIPTION:
TB is an infectious disease caused by the bacillus Mycobacterium tuberculosis. It typically affects the lungs (pulmonary TB) but can also affect other sites (extrapulmonary TB). The disease is spread when people who are sick with pulmonary TB expel bacteria into the air, for example by coughing. Overall, a relatively small proportion (5-15%) of the estimated 1.7 billion people infected with M. tuberculosis will develop TB disease (active disease) during their lifetime. However, the probability of developing TB disease is much higher among people infected with HIV, and also higher among people affected by risk factors such as under-nutrition, diabetes, smoking and alcohol consumption. Latent tuberculosis infection (LTBI) is defined as a state of persistent immune response to stimulation by Mycobacterium tuberculosis antigens with no evidence of clinically manifest active TB. As there is no "gold standard" test for LTBI, the global burden is not known with certainty; however, up to one third of the world's population is estimated to be infected with M. tuberculosis , and the vast majority have no signs or symptoms of TB disease and are not infectious, although they are at risk for active TB disease and for becoming infectious. Several studies have shown that, on average, 5-10% of those infected will develop active TB disease over the course of their lives, usually within the first 5 years after initial infection . The risk for active TB disease after infection depends on several factors, the most important being immunological status

ELIGIBILITY:
Inclusion Criteria:

children aged under 5 yearsold with one of the following risk factor :

1. have diabetes
2. have chronic kidney disease or receive haemodialysis

Exclusion Criteria:

1. All children aged above 12 years old
2. History of recent contact with TB positive patient
3. All children under 5 yearsold without any other risk factor

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients without active TB sequelae in their CXR
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Latent Tuberculosis in High Risk Young Children Attending Pediatric Hospital of Assiut University | one year
  To identify the prevalence of latent tuberculosis (according to new guideline ;NICE tuberculosis) among these high risk groups of children and notify ministry of health

CONTACTS AND LOCATIONS:
Overall Officials: nagla h. fargaly, professor, Study Director — Assiut University

REFERENCES:
- [Background] Getahun H, Matteelli A, Chaisson RE, Raviglione M. Latent Mycobacterium tuberculosis infection. N Engl J Med. 2015 May 28;372(22):2127-35. doi: 10.1056/NEJMra1405427. No abstract available. PMID 26017823
- [Background] Corbett EL, Watt CJ, Walker N, Maher D, Williams BG, Raviglione MC, Dye C. The growing burden of tuberculosis: global trends and interactions with the HIV epidemic. Arch Intern Med. 2003 May 12;163(9):1009-21. doi: 10.1001/archinte.163.9.1009. PMID 12742798
- [Background] Comstock GW, Livesay VT, Woolpert SF. The prognosis of a positive tuberculin reaction in childhood and adolescence. Am J Epidemiol. 1974 Feb;99(2):131-8. doi: 10.1093/oxfordjournals.aje.a121593. No abstract available. PMID 4810628